CLINICAL TRIAL: NCT03396588
Title: Non-Opiate Treatment After Prenatal Opiate Exposure to Prevent Postnatal Injury to the Young Brain
Acronym: No-POPPY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henrietta Bada (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Henrietta Bada, Professor of Pediatrics, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-0534-F34; 1R01DA043519-01 (NIH)
Record Dates: First submitted 2017-12-13; First posted 2018-01-11 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Opiate use during pregnancy; Clonidine; Morphine; Prenatal opiate; Neonatal Abstinence Syndrome; Infant, Newborn, Diseases; Substance-Related Disorders; Chemically-Induced Disorders; Opiate Alkaloids; Mental Disorders; Narcotics; Central Nervous System Depressants; Physiological Effects of Drugs; Adrenergic alpha-2 Receptor Agonists; Adrenergic alpha-Agonists; Molecular Mechanisms of Pharmacological Action; Antihypertensive Agents; Analgesics; Peripheral Nervous System Agents; Sympatholytics; Autonomic Agents; Neurotransmitter Agents
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Infant, Newborn, Diseases; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders | interventions — Clonidine; Morphine

STUDY DESIGN:
Intervention Model Description: The study is intended to treat NAS using a randomized and double-blind study design to compare the use of opiate (morphine) or non-opiate (clonidine). Newborns meeting the study criteria for drug withdrawal and treatment will be randomized to receive one of the drugs (morphine, clonidine). Newborns requiring a second drug to help relieve the symptoms will be treated with phenobarbital for both groups. Randomization, blinding and dispensing will occur in the Investigational Drug Services Unit. Nursing personnel in the NICU will be masked to the treatment administered to each baby.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will mask parents and child caregivers, and NICU nurses giving the drug, other personnel, residents and attending physicians, and research staff. Since initial dose is set using weight based-dosing, a physician's order can be entered in the electronic medical record to give the initial study drug with the infant's weight stated in the order. Increase in dosing will be ordered as to increase by 25% of initial dose or decrease of dose by 10% of maximum dose. During the pilot study, masking of treating personnel was maintained while the hospital pharmacist was the only person aware of which study drug the infant was receiving. The examiners for administration of the NNNS and the research nurse and research case worker will be masked to treatment received. Those seeing the infant in the clinic will also be masked to the treatment assignment. Morphine and clonidine are dispensed in identical appearance, color, smell, and volume.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clonidine (Active Comparator): Babies randomized to clonidine will receive 1mcg/kg/dose (with a dosing interval of 3 or 4 hours).
  Interventions: Drug: Clonidine
- Morphine (Active Comparator): Babies randomized to morphine will receive 0.06 mg/kg/dose (with a dosing interval of 3 or 4 hours).
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Clonidine — 1mcg/kg/dose (with a dosing interval of 3 or 4 hours), increases by 25% of initial dose every 12-24 hrs. Decrease by 10% of max dose every 24 hrs.
  Other Names: clonidine hydrochloride
  Arms: Clonidine
Drug: Morphine — Starting dose is 0.06 mg/kg/dose (every 3 or 4 hours), increases by 25% of initial dose every 12-24 hrs. Decrease by 10% of max dose every 24 hrs.
  Other Names: Morphine Sulfate
  Arms: Morphine

SUMMARY:
The long term goals of our research are to establish the best pharmacological treatment for NAS and determine how pharmacologic treatment of NAS affects long-term developmental outcomes. The objective of this application is to evaluate the effectiveness of clonidine as a treatment for neonates with NAS, in a randomized clinical trial. Our central hypothesis is that clonidine will effectively treat drug withdrawal manifestations in neonates.

DETAILED DESCRIPTION:
In this current proposal, the research plan is based on our pilot study, which randomized infants with NAS to receive morphine or clonidine. The treatment groups were similar as to mean birth weight, gestational age, Apgar scores, and postnatal age at treatment. Infants enrolled had no other medical or surgical complications. Treatment was initiated per our NICU standard at the time, and will be continued in this protocol. Total LOS was shorter by about 1 week in the clonidine (mean of 15 days), compared to 21 days in the morphine group.

Aims and Objectives:

To determine whether the treatment of NAS with a non-opiate medication, clonidine, will be more effective than morphine

* Compare Clonidine and morphine for the treatment of NAS. Compare the efficacy of each drug which is determined by duration of treatment in number of days, number of dose escalations needed to achieve needed treatment, and the need for second drug treatment.
* Evaluate the neurobehavioral performance scores (habituation, orientation, self- regulation, motor/reflexes, and stress/ abstinence scales) using the neonatal intensive care (NICU) network neurobehavioral scale (NNNS) in both treatment groups. This exam will take place after treatment begins, and at one month post-natal age (38-44 weeks post menstrual age) or at discharge, whichever comes first.

To determine whether treatment of NAS with clonidine will result in better early childhood outcomes than those treated with morphine • Compare the cognitive, motor and behavioral development of children in both treatment groups using the Bayley III Scales of Infant Development at 6 months, one and two years of age.

To build population pharmacokinetic/pharmacodynamic models and determine factors that affect exposure and response to morphine and clonidine

• Measure blood levels obtained at random times and correlate to Finnegan scores. The pharmacodynamics may help with understanding NAS medications and coping measures in babies.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) > or equal to 35 weeks
* Known prenatal opiate exposure (by mother admitting use, mom with positive opiate screen during pregnancy, or positive neonatal urine and meconium screening)
* No known prenatal cocaine exposure
* No morphine or clonidine dose before enrollment
* Symptomatic with Finnegan scores (FS): 3 consecutive scores greater than or equal to 8, OR 2 consecutive scores greater than or equal to 12, and/or with attending decision to treat for NAS
* Less than or equal to 7 days of age
* Attending physician decides to start pharmacologic treatment and agrees to infant's study participation

Exclusion Criteria:

* Seizures
* Major congenital malformations
* Blood pressure instability
* Major medical condition in addition to NAS
* Parents unable to understand English

Ages: 12 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrietta S Bada, MD MPH, Principal Investigator — University of Kentucky
Locations (1):
- Kentucky Children's Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bada HS, Sithisarn T, Gibson J, Garlitz K, Caldwell R, Capilouto G, Li Y, Leggas M, Breheny P. Morphine versus clonidine for neonatal abstinence syndrome. Pediatrics. 2015 Feb;135(2):e383-91. doi: 10.1542/peds.2014-2377. PMID 25624389
- [Background] Lester BM, Tronick EZ, LaGasse L, Seifer R, Bauer CR, Shankaran S, Bada HS, Wright LL, Smeriglio VL, Lu J. Summary statistics of neonatal intensive care unit network neurobehavioral scale scores from the maternal lifestyle study: a quasinormative sample. Pediatrics. 2004 Mar;113(3 Pt 2):668-75. PMID 14993525

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clonidine | Morphine
Started | 60 | 60
Completed | 58 | 57
Not Completed | 2 | 3
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine | Morphine | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 60 | 120
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] — gestational age
  weeks | 38.7 (1.2) | 38.3 (1.3) | 38.4 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 37 | 30 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 60 | 56 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 53 | 52 | 105
  More than one race | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurobehavioral Performance Summary Scores From the Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS)
Description: The summary scores from the Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) give a measure of infant neurobehavior in the following areas (score range): habituation (1-9), regulation (2.20-7.50), attention (1.29-8.4), Handling (0-1), quality of movement (1.20-6.20), Non-optimal reflexes (0-12), Asymmetric reflexes (0-7), arousal (2.43-6.67), hypertonicity (0-8), hypotonicity (0-5.0), excitability (0-11), lethargy (0-11.0), and stress/abstinence (0-0.57). A higher score for each item means a higher level of the construct. For example, a higher score for hypertonicity means the infant is more hypertonic and higher score on hypotonicity means the infant is more hypotonic. No cut-off score published for normal or abnormal behavioral performance.
Time Frame: Baseline (5-10 days post natal age) and one-month post-natal age (between 4-6 weeks of age), or at discharge, whichever comes first.
Population: Some babies were unable to be assessed in certain domains and therefore were not included in the total analyzed for that domain.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 54 | 51
score on a scale
  Habituation: number analyzed (Participants) | 9 | 15
  Habituation | 0.5 [-1.0 to 1.0] | 0.3 [-1.0 to 1.0]
  Attention: number analyzed (Participants) | 31 | 31
  Attention | 1.0 [-0.1 to 2.0] | 0.6 [0.2 to 1.6]
  Handling: number analyzed (Participants) | 35 | 37
  Handling | -0.1 [-0.4 to 0.1] | 0.1 [0.0 to 0.4]
  Quality of movement: number analyzed (Participants) | 52 | 51
  Quality of movement | 0.1 [-0.3 to 0.8] | 0.0 [-0.5 to 0.5]
  Regulation: number analyzed (Participants) | 52 | 51
  Regulation | 0.5 [-0.5 to 1.3] | -0.2 [-0.8 to 0.2]
  Non-optimal reflexes | -1.0 [-2.5 to 1.0] | -1.0 [-2.0 to 1.0]
  Asymmetry total/reflexes | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Arousal | -0.1 [-0.6 to 0.3] | 0.4 [0.0 to 0.7]
  Hypertonia | -1.0 [-2.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Hypotonia | 0.0 [0.0 to 0.5] | 0.0 [0.0 to 0.0]
  Excitability | -1.0 [-3.0 to 1.0] | 1.0 [-1.0 to 3.0]
  Lethargy | 0.0 [-0.1 to 0.0] | 0.0 [0.0 to 0.1]
  Stress abstinence | 0.0 [-0.1 to 0.0] | 0.0 [0.0 to 0.1]

2. Primary Outcome: Bayley Scales of Infant and Toddler Development Third Edition
Description: Scores obtained Bayley Scales of Infant and Toddler Development Third Edition in the developmental domains of motor, cognitive, and language. This tool for measures of motor, cognitive, and language development is a series of standardized measurements and for each domain, the standardized scores have a mean of 100 and standard deviation of 15 with a range of 55-155 for cognitive and a range of 45-155 for language and motor (lower scores indicating greater impairment). Scores below 1 standard deviation (=or less than 84) is considered below normal. Scores above 1 standard deviation (over 115) represent higher than normal functioning in each domain. The score for each domain (motor, cognitive, and language functioning) represents the composite score.
Time Frame: 6 months of life
Population: Participants may not have had the 6 month Bayley due to the participant being lost to follow up, or because of COVID-19 research restrictions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 32 | 38
score on a scale
  Cognitive | 113.0 (12.8) | 111.8 (11.1)
  Language | 91.8 (13.4) | 87.7 (13.5)
  Motor | 102.4 (16.4) | 97.4 (12.3)

3. Primary Outcome: Bayley Scales of Infant and Toddler Development Third Edition
Description: as for outcome 2
Time Frame: 1 year of life
Population: Participants may not have had the 12 month Bayley due to the participant being lost to follow up, or because of COVID-19 research restrictions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 19 | 18
score on a scale
  Cognitive | 98.2 (11.5) | 97.2 (10.8)
  Language | 91.8 (11.6) | 92.2 (12.2)
  Motor | 99.1 (12.2) | 96.2 (9.3)

4. Primary Outcome: Bayley Scales of Infant and Toddler Development Third Edition
Description: as for outcome 2
Time Frame: 2 years of life
Population: Participants may not have had the 24 month Bayley due to the participant being lost to follow up, or because of COVID-19 research restrictions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 7 | 8
score on a scale
  Cognitive | 84.3 (6.7) | 81.1 (9.6)
  Language | 95.4 (9.4) | 86.2 (11.0)
  Motor | 97.6 (7.2) | 96.0 (9.8)

5. Primary Outcome: Ages and Stages Questionnaire Third Edition (ASQ-3)
Description: The ASQ-3 is a developmental screening tool to assess developmental progress in children. Children are scored in the areas of communication, gross motor skills, fine motor skills, problem solving, and personal/social skills. The child's parent/guardian answers whether their child already does an activity (yes=10), sometimes does it (sometimes=5), or does not yet do it (not yet=0). The answers are then used to score each category. Each category is then broken down into whether the child falls above the cutoff (child development is on schedule), close to the cutoff (child development is slightly delayed and requires monitoring/intervention), or below the cutoff (delayed development and further assessment required).
Time Frame: 12 months of age
Population: ASQ-3 assessments were used for babies who were unable to have Bayley assessment performed due to COVID-19 research restrictions. The babies who had the Bayley did not have the ASQ.
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 7 | 10
Participants
  Communication: Above cutoffs | 6 | 7
  Communication: Close to cutoffs | 0 | 3
  Communication: Below cutoffs | 1 | 0
  Gross motor: Above cutoffs | 7 | 10
  Gross motor: Close to cutoffs | 0 | 0
  Gross motor: Below cutoffs | 0 | 0
  Fine motor: Above cutoffs | 6 | 8
  Fine motor: Close to cutoffs | 1 | 2
  Fine motor: Below cutoffs | 0 | 0
  Problem solving: Above cutoffs | 4 | 9
  Problem solving: Close to cutoffs | 3 | 1
  Problem solving: Below cutoffs | 0 | 0
  Personal/social: Above cutoffs | 7 | 10
  Personal/social: Close to cutoffs | 0 | 0
  Personal/social: Below cutoffs | 0 | 0

6. Primary Outcome: Ages and Stages Questionnaire Third Edition (ASQ-3)
Description: as for outcome 5
Time Frame: 24 months
Population: The ASQ-3 at 24 months was used for babies who were unable to have the Bayley assessment due to COVID-19 research restrictions.
  The babies who had the Bayley did not have the ASQ performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 14 | 11
Participants
  Communication: Above cutoffs | 8 | 8
  Communication: Close to cutoffs | 2 | 2
  Communication: Below cutoffs | 4 | 1
  Gross motor: Above cutoffs | 13 | 10
  Gross motor: Close to cutoffs | 1 | 1
  Gross motor: Below cutoffs | 0 | 0
  Fine motor: Above cutoffs | 8 | 8
  Fine motor: Close to cutoffs | 4 | 3
  Fine motor: Below cutoffs | 2 | 0
  Problem solving: Above cutoffs | 12 | 9
  Problem solving: Close to cutoffs | 2 | 2
  Problem solving: Below cutoffs | 0 | 0
  Personal/social: Above cutoffs | 12 | 10
  Personal/social: Close to cutoffs | 1 | 1
  Personal/social: Below cutoffs | 1 | 0

7. Primary Outcome: Childhood Behavior Checklist (CBCL) T-Scores
Description: The CBCL/1.5-5 is validated for children ages 1.5 to 5 years old. It obtains caregivers' ratings of 113 behavior items.
  Scores are broken down into internalizing problems (scores range 29-100, normal is below 60), externalizing problems (scores range from 28-100, normal is below 60), and total problems (range is 28-100, normal is below 60).
  Items are scored on the following syndrome scales: Emotionally Reactive, Anxious/Depressed, Somatic Complaints, Withdrawn, Attention Problems, Aggressive Behavior, and Sleep Problems. Items are also scored on the following DSM-oriented scales: Affective Problems, Anxiety Problems, Pervasive Developmental Problems, Attention Deficit/Hyperactivity Problems, Stress Problems, Autism Spectrum Problems, and Oppositional Defiant Problems.
  The CBCL consists of 113 items, scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often)
Time Frame: Once post discharge (between 18 months up to 24 months of age)
Population: Only children in the treated cohorts had the CBCL.
  Participants who were considered lost to follow up did not have the CBCL.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 15 | 24
score on a scale
  Internalizing Problems | 52.31 (10.4) | 50.9 (13.9)
  Externalizing Problems | 54.8 (13.4) | 53.5 (17.0)
  Total Problems | 53.6 (12.6) | 53.5 (13.5)

8. Secondary Outcome: Duration of Treatment
Description: Total number days of treatment
Time Frame: 60 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 60 | 60
days | 17 [15 to 19] | 15 [13 to 17]

9. Secondary Outcome: Childhood Behavior Checklist 1.5-5 T-Scores
Description: On the CBCL 1.5-5, T-scores, with a mean of 50 and a standard deviation of 10, are used to interpret results, with scores of 65 or higher indicating a clinical range, and scores between 60 and 64 suggesting a borderline clinical range.
Time Frame: Once post discharge (between 18 months up to 24 months of age)
Population: Participants who were lost to follow up did not have the CBCL.
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Morphine
Number analyzed (Participants) | 15 | 24
Participants
  Internalizing Problems Borderline T-Scores | 5 | 2
  Internalizing Problems Clinical Range T-Scores | 1 | 8
  Externalizing Problems Borderline T-Scores | 2 | 2
  Externalizing Problems Clinical Range T-Scores | 3 | 6
  Total Problems Borderline T-Scores | 3 | 2
  Total Problems Clinical Range T-Scores | 1 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent until the subject was off study. For subjects who completed the entire study, the maximum amount of time for AE collection is 26 months from date of consent.
Description: AEs were collected through the health system EMR and patient reports.
Arm/Group | Clonidine | Morphine
All-Cause Mortality (participants affected / at risk) | 1/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 9/60 | 15/60
Other Adverse Events (participants affected / at risk) | 52/60 | 24/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clonidine (N=60) | Morphine (N=60)
Sustained tachycardia (Cardiac disorders) | 3 | 4 — >180 BPM for at least 3 hours
Skin lesions (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperthermia (General disorders) | 0 | 1
Respiratory Distress (Reproductive system and breast disorders) | 1 | 1
Increased Heart Rate (Cardiac disorders) | 1 | 0
Hematochezia (Gastrointestinal disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 4 | 1
Seizure (Nervous system disorders) | 0 | 2
Respiratory Syncytial Virus (Infections and infestations) | 0 | 2
Hypothermia (General disorders) | 1 | 1
Dehydration (Gastrointestinal disorders) | 1 | 0
Poor feeding (General disorders) | 0 | 2
Pyloric stenosis (Gastrointestinal disorders) | 0 | 2
Undescended testicle (Renal and urinary disorders) | 0 | 1
Persistent ear infections (Ear and labyrinth disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clonidine (N=60) | Morphine (N=60)
Finnegan scores consecutively >8 (Nervous system disorders) | 24 | 17
Adjunct medication added (Investigations) | 13 | 2
Phenobarbitol added (Investigations) | 15 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03396588/Prot_SAP_ICF_002.pdf